CLINICAL TRIAL: NCT00639145
Title: Maternal Events and Pregnancy Outcomes in a Cohort of Human Immunodeficiency Virus-Infected Women Receiving Antiretroviral Therapy in Sub- Saharan Africa
Brief Title: Elizabeth Glaser Pediatric AIDS Foundation Maternal Events and Pregnancy Outcomes (MEP Project)A Multi-site Protocol
Acronym: MEPProject
Status: Completed | Type: Observational
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Centre for Infectious Disease Research in Zambia (CIDRZ) (Unknown); University of Limpopo MEDUNSA (Unknown); Health Systems Trust (Other)
Responsible Party: Sponsor
Other Study IDs: EG001
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: HIV Infections; HIV Positive; Pregnant Women
Keywords: HIV; Pregnancy; Antiretrovirals; HIV Seronegativity; Treatment Experienced
MeSH Terms: conditions — HIV Infections; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find out if antiretroviral drugs are safe and well tolerated by HIV-positive pregnant women and their infants in South Africa and Zambia.

DETAILED DESCRIPTION:
Although the use of HAART in pregnancy has significantly reduced rates of vertical transmission of HIV-1, some questions remain regarding the safety of these therapies and their potential impact on the uninfected infant.

The overall goal of the project is to establish a voluntary exposure-registry and perform observational surveillance on HIV - positive pregnant women who are exposed to antiretroviral products during the prenatal period, in order to evaluate the outcome of the pregnancy and safety of the products in HIV-positive pregnant women, and their infants.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive pregnant woman on antiretroviral treatment
* Able and willing to participate and provide informed consent
* Be at least 18 years of age or older than legal age to provide consent
* If under legal age, must have legal guardian who is able to give consent
* Be an emancipated minor

Exclusion Criteria:

* History of mental illness
* History of condition that would preclude provision of consent
* Inability to provide consent

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV positive pregnant women attending ART clinics
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of Congenital birth defects | At birth
  Number of congenital birth defects among infants born in the study

SECONDARY OUTCOMES:
Adverse Pregnancy outcomes | At outcome of pregnancy
  Pregnancy outcomes other than normal live birth such as preterm birth, stillbirth and low birth weight

CONTACTS AND LOCATIONS:
Overall Officials: Richard Marlink, MD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (2):
- University of Limpopo / Elizabeth Glaser Pediatric AIDS Foundation, Medunsa, South Africa
- Center for Infectious Disease Research in Zambia (CIDRZ), Lusaka, Zambia